CLINICAL TRIAL: NCT07222605
Title: Research Study Evaluating Patient Experience With the MemorEM for Patients With Neurological Diseases
Brief Title: Research Study for Patients With Neurological Diseases Which Evaluates the Patient Experience of the MemorEM Device
Acronym: MemorEM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: eQ8Health Corporation d/b/a CareONE Concierge (Industry)
Collaborators: NeuroEM Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CareONE-002
Record Dates: First submitted 2025-07-08; First posted 2025-10-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Parkinson Disease; Frontotemporal Dementia; Cortico Basal Degeneration; Posterior Cortical Atrophy (PCA); Neurological Diseases or Conditions; Dementia
Keywords: Alzheimer; Dementia; Cognitive Impairment; FDA Breakthrough Device
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Frontotemporal Dementia; Corticobasal Degeneration; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patient Experience Arm (Active Comparator)
  Interventions: Device: MemorEM

INTERVENTIONS:
Device: MemorEM — The MemorEM device delivers 915MHz electromagnetic waves to the head via emitters in a cap worn on the head and powered by a control box and battery worn on the arm.

SUMMARY:
Primary Objective:

The primary objective of this pilot study is to gain voluntary feedback from patients with neurological diseases and their caregivers regarding their experiences using the MemorEM head device. This information may help in new designs of the MemorEM and suggest ways to increase compliance for future clinical trials and eventual commercialization.

Secondary Objective:

The secondary objective is to note areas of potential improvement in the progression of the subject's neurological disease and identify the potential for the MemorEM to treat neurological diseases other than Alzheimer's disease. The investigators are also interested in Alzheimer's variants like those with ApoE4 alleles (none of the participants in the 8-person pilot were Apo-E4 positive), known mutations causing early onset Alzheimer's, and Posterior Cortical Atrophy.

DETAILED DESCRIPTION:
Study Duration:

The study will be open-ended with patients continuing use of the MemorEM as they wish or when NeuroEM Therapeutics recalls the device. It is expected but optional that patients will use the devices for approximately two years.

Study Design:

This study will focus on the "patient experience" of using the MemorEM device over an extended time period. Patients will remain under the care of their physicians and will provide brief descriptions of their device experiences and any suggestions for improvements. This study will not require any interventions other than using the MemorEM device, which was rated as Non-Significant Risk by the Western IRB for the previous pilot trial including two extensions that raised no safety concerns over the two and a half years of treatment.

Study Population:

The study population will consist of various patients suffering from diagnosed neurological diseases. Patients may be selected from those diagnosed with Alzheimer's disease, Frontotemporal dementia, Posterior cortical atrophy, Corticobasal dementia, Parkinson's disease, and other neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a neurological disease involving aggregated proteins such as Alzheimer's and its variants, Parkinson's, Frontotemporal dementia, Amyotrophic lateral sclerosis, Tauopathies, and other related neurological diseases.
* Presence of a caregiver(s) responsible for ensuring treatment compliance and potentially with authority to make medical decisions for the patient if the patient is not competent to make those decisions.
* A statement from each patient's physician that indicates the patient has the ability to understand and consent on their own AND they have the willingness to sign CareONE's patient consent.

Exclusion Criteria:

* Patient has Seizures, Epilepsy, uncontrolled Depression, uncontrolled Bipolar disorder, psychotic disorders, alcoholism or drug addiction
* Presence of metal implants in the head, except for metal dental implants
* Patient has hypertension that is unresponsive to anti-hypertensive medications
* Patient has implanted medication pumps unless cleared by physician
* Patient has significant heart disease, as determined by a physician

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient and caregiver reports on device design and use | Surveys will be given starting a month after beginning treatment and monthly thereafter over the course of up to two years.
  The primary objective of this pilot study is to gain voluntary feedback from patients with neurological diseases and their caregivers regarding their experiences using the MemorEM head device. This information will be gathered via a monthly survey. This information may help in new designs of the MemorEM and suggest ways to increase compliance for future clinical trials and eventual commercialization.

SECONDARY OUTCOMES:
Reports of efficacy in treating a patient's neurological condition | Surveys will be given starting a month after beginning treatment and monthly thereafter over the course of up to two years.
  The secondary objective is to note areas of potential improvement in the progression of the subject's neurological disease and identify the potential for the MemorEM to treat neurological diseases other than Alzheimer's disease. The investigators are also interested in Alzheimer's variants like those with ApoE4 alleles, known mutations causing early onset Alzheimer's, and Posterior Cortical Atrophy. The monthly survey contains questions designed to identify changes in cognition, mood, physical symptoms, activities of daily living, and capture any narrative information provided by patient or caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Cavolina, PharmD, Principal Investigator — Principal Investigator
Locations (1):
- CareONE Concierge, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share all study results (de-identified) with study collaborator (NeuroEM)
Supporting Information: Study Protocol, ICF
Time Frame: Dec 2025 for each contiguous month through the end of the first phase of the study which is Dec 2026.
Access Criteria: The Principal Investigator (Edward Goodwin, PharmD) of NeuroEM will be the recipient of IPD
URL: https://www.neuroem.com